CLINICAL TRIAL: NCT06070402
Title: Use of a Voice Assistant (DIAL) to Improve Unwanted Loneliness, Mental Health, and Quality of Life in Older People: a Randomized Controlled Trial
Brief Title: Use of a Voice Assistant to Improve Mental Health in Older People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Valencia (Other)
Collaborators: Universitat Politècnica de València (Other); Iniciativa Social Integral (Unknown); Las Naves (Unknown)
Responsible Party: Principal Investigator, Rosa M. Baños Rivera, Principal Investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1828511
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Depression; Loneliness; Anxiety; Quality of Life
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Experimental design with two groups: the control group and the experimental group, using pre and post evaluations by means of a randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants randomly assigned to this group will test the DIAL device for four weeks
  Interventions: Device: DIAL, a voice-controlled virtual assistant
- Control group (No Intervention): Participants randomly assigned to this group will not use the DIAL device

INTERVENTIONS:
Device: DIAL, a voice-controlled virtual assistant — Participants in the experimental group will test in their homes a device called DIAL, a voice-controlled virtual assistant designed to communicate with the elderly and help them in different contexts. They will use it for four weeks. They will receive an individual training session on how to use the device, an instruction sheet for its use and, in addition, they will receive telephone technical support throughout the study. Finally, the device will be uninstalled and all participants will be called back to answer the same survey they answered before the intervention.
  Arms: Experimental group

SUMMARY:
The main objective of this study is to evaluate the effectiveness of DIAL (an innovative and user-friendly solution based on Multiplatform Voice Assistive Technologies) in reducing unwanted loneliness and increasing the mental health and the quality of life in individuals over 65 years old. Additionally, a secondary objective is to evaluate the experience of using the system, including aspects of usability and satisfaction, and to analyze whether the functionalities provided by DIAL contribute to the improvement of various dimensions in the lives of the elderly. It is hypothesized that DIAL will reduce unwanted loneliness and improve mental health in older people. In addition, we aim to obtain positive ratings in terms of usability and satisfaction with DIAL, along with the verification that most of the functionalities provided by DIAL will be useful to older people.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the effectiveness of DIAL in reducing unwanted loneliness and increasing the mental health and the quality of life of elderly people. Additionally, a secondary objective is to evaluate the experience of using the system, including aspects of usability and satisfaction, and to analyze whether the functionalities provided by DIAL contribute to the improvement of various dimensions in the lives of the elderly. For this purposes, a randomized controlled trial with a control group and an experimental group will be conducted in Valencia at the end of 2023. Participants in the experimental group will use DIAL for four weeks. All participants will complete different measures of mental health and quality of life, as well as measures related to the experience of using DIAL. Mixed ANOVA tests will be used to determine if there were statistically significant differences between the different measures evaluated. An alpha of 0.05 will be taken as the confidence level. In addition, a descriptive study will be conducted on the variables related to the DIAL user experience. It is hypothesized that DIAL will reduce unwanted loneliness and improve mental health in older people. In addition, we aim to obtain positive ratings in terms of usability and satisfaction with DIAL, along with the verification that most of the functionalities provided by DIAL will be useful to older people.

ELIGIBILITY:
Inclusion Criteria:

* 1) Be 65 years old or older, 2) Speak Spanish, 3) Meet at least one criterion of vulnerability to suffering unwanted loneliness (the criteria will be taken from the European report by Baarck et al. 2021. For example, being a widower, have a physical illness...), 4) Ability and willingness to participate in the study.

Exclusion Criteria:

* 1) Present cognitive impairment, 2) Suffer from a serious mental problem (e.g. depression, schizophrenia) or 3) Suffer from a serious physical problem (e.g. blindness or deafness) that makes interaction with the device difficult.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-11-15 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale (UCLA; Russell et al., 1980; Vázquez & Jiménez, 1994) | Pre-intervention, immediately after the intervention, and follow-up (3 months)
  The instrument measures the feeling of loneliness and consists of 20 items, 11 of which are negative (for example, I lack company) and nine positive (for example, I feel in tune with the people around me). All items are scored from 1 (never) to 4 (frequently). After reversing the score on items 1, 5, 6, 9, 10, 15, 16, 19 and 20, the scores corresponding to the 20 items are added, obtaining a total isolation score. The range of scores goes from 20 to 80, with a higher score corresponding to a greater degree of loneliness
Health-related quality of life scale (EuroQol-5D; Herdman et al., 2001). | Pre-intervention, immediately after the intervention, and follow-up (3 months)
  This scale measures five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each category consists of 1 item, ranging from 1 (no problems) to 3 (many problems). The second part of the EQ-5D-3L is a 20-centimeter vertical visual analog scale, ranging from 0 (worst imaginable health state) to 100 (best imaginable health state). The individual must mark the point on the scale that best reflects the assessment of their current global health status. The use of the VAS provides a complementary score to the descriptive system of self-assessment of the individual's health status
The World Health Organization Quality of Life-Old (WHOQOL-OLD Scale; Power et al., 2005; Lucas-Carrasco et al., 2011). | Pre-intervention, immediately after the intervention, and follow-up (3 months)
  The WHOQOL-OLD is a 24-item self-report instrument that is divided into six facets: Facet 1- Sensory abilities (items 1, 2, 10, 20); Facet 2- Autonomy (items 3, 4, 5, 11); Facet 3- Past, present and future activities (items 12, 13, 15, 19); Facet 4- Social participation (items 14, 16, 17, 18); Facet 5- Death (items 6, 7, 8, 9); and Facet 6- Intimacy (items 21, 22, 23, 24). Responses are based on a 5-point Likert-type response scale (ranging from 1-5), with items 1, 2, 6, 7, 8, 9, and 10 reverse scored. WHOQOL-OLD total scores in each facet range from 4 to 20, with higher scores indicating better quality of life. A global score (general QOL - GQOL) is also calculated from the set of 24 items
The Generalized Anxiety Disorder Questionnaire-2 (GAD-2; Kroenke et al., 2007; García-Campayo et al., 2012) | Pre-intervention, immediately after the intervention, and follow-up (3 months)
  It is a self-report measure containing 2 items assessing anxiety symptoms. The items are scored on a 4-point Likert scale, ranging from 0 (no days) to 3 (almost every day), where a high score indicates greater anxiety symptoms
The Patient Health Questionnaire-2 (PHQ-2; Kroenke et al., 2003; Rodríguez-Muñoz et al., 2017) | Pre-intervention, immediately after the intervention, and follow-up (3 months)
  It is a self-report measure consisting of 2 items assessing depressive symptoms. The items are scored on a 4-point Likert scale, ranging from 0 (never) to 3 (almost every day), where a high score indicates higher levels of depressive symptoms

SECONDARY OUTCOMES:
The System Usability Scale (SUS; Brooke, 1996; Sevilla González et al., 2020) | Immediately after the intervention
  It is a self-reported measure that assesses the overall usability of the tool. It is a 10-item scale, measured on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Total SUS scores range from 0 to 100.The questionnaire is designed to be answered after the user's interaction with the system
The Client Satisfaction Questionnaire (CSQ; Roberts & Attkisson, 1983) | Immediately after the intervention
  It is a self-report questionnaire that assesses the patient's overall satisfaction with the tool. It consists of 8 items on a 4-point Likert scale ranging from 1 (lowest score per item) to 4 (highest score per item). The total score ranges from 8 to 32, with higher values indicating higher satisfaction
Price they would be willing to pay | Immediately after the intervention
  We will ask them what price they would be willing to pay for DIAL, between 0 and 100 euros per month
Questions about skills | Immediately after the intervention
  Older people will be asked if DIAL has helped them in different facets of their lives. Specifically, if it has helped them to: improve their mood, feel more understood, feel listened to, feel supported, feel more supported, feel more accompanied, drink more water, have better hygiene, walk more, take their medication better, move more, talk more with people close to them, be more in contact with people close to them (family or friends)
Aspects related to the DIAL voice assistant | Immediately after the intervention
  They will be asked what aspects have improved in their life since the application has been installed in their home
Aspects related to DIAL's complementary care services (support person) | Immediately after the intervention
  They will be asked what aspects have improved in their life since they have had the complementary services of DIAL (the support person)

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Mª Baños, Full professor, Principal Investigator — University of Valencia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol